CLINICAL TRIAL: NCT05351827
Title: Mild Intermittent Hypoxia: A Prophylactic for Autonomic Dysfunction in Individuals With Spinal Cord Injuries
Acronym: MIH and AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: John D. Dingell VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3847-W; IRB-22-04-4550 (Other: John D. Dingell VA Medical Center)
Record Dates: First submitted 2022-04-18; First posted 2022-04-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Autonomic Dysreflexia
MeSH Terms: conditions — Spinal Cord Injuries; Autonomic Dysreflexia | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mild Intermittent Hypoxia (Experimental): This arm of the protocol will receive mild intermittent hypoxia (8% Oxygen) with end-tidal carbon dioxide maintained 1-3 millimeters of mercury above baseline, while in the laboratory. If diagnosed with sleep apnea, participants will be treated with continuous positive airway pressure for the duration of the intervention.
  Interventions: Other: Mild Intermittent Hypoxia
- Sham (Sham Comparator): This arm of the protocol will receive sham air (21 % Oxygen) while in the laboratory. No additional gases will be employed. If diagnosed with sleep apnea, participants will be treated with continuous positive airway pressure for the duration of the intervention.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Mild Intermittent Hypoxia — Participants will breathe 8% oxygen through a non-diffusable bag that is connected to a 5-way stopcock. The inspiration side of the system is then connected to a 2-way non-rebreathing valve which is connected to a pneumotachometer that is connected to a tight fitting facemask. 100% oxygen and carbon dioxide are titrated into the system to ensure the appropriate hypoxic and hypercapnic stimulus is delivered. The investigators will lower oxygen to 55-60 mmHg and maintain end-tidal carbon dioxide 1-3 mmHg above individual baseline values. The protocol starts with 10 minutes of baseline breathing (room air) then followed by 10 more minutes of breathing room air with the additional carbon dioxide. Thereafter, individuals undergo 12 2-minute bouts of hypoxia with 2 minutes of normoxia (room air) interspersed between episodes. The intervention protocol concludes with 20 minutes of monitoring all breathing and cardiovascular measurements.
  Arms: Mild Intermittent Hypoxia
Other: Sham — Participants will breathe 21% oxygen through a non-diffusable bag that is connected to a 5-way stopcock. The inspiration side of the system is then connected to a 2-way non-rebreathing valve which is connected to a pneumotachometer that is connected to a tight fitting facemask. No supplemental oxygen or carbon dioxide will be used during the sham protocol. The protocol starts with 10 minutes of baseline breathing (room air) then followed by 10 more minutes of breathing room air with the additional carbon dioxide. Thereafter, individuals undergo 12 2-minute bouts of hypoxia with 2 minutes of normoxia (room air) interspersed between episodes. The intervention protocol concludes with 20 minutes of monitoring all breathing and cardiovascular measurements.
  Arms: Sham

SUMMARY:
The prevalence of autonomic dysfunction and sleep disordered breathing (SDB) is increased in individuals with spinal cord injury (SCI). The loss of autonomic control results in autonomic dysreflexia (AD) and orthostatic hypotension (OH) which explains the increase in cardiovascular related mortality in these Veterans. There is no effective prophylaxis for autonomic dysfunction. The lack of prophylactic treatment for autonomic dysfunction, and no best clinical practices for SDB in SCI, are significant health concerns for Veterans with SCI. Therefore, the investigators will investigate the effectiveness of mild intermittent hypoxia (MIH) as a prophylactic for autonomic dysfunction in patients with SCI. The investigators propose that MIH targets several mechanisms associated with autonomic control and the co-morbidities associated with SDB. Specifically, exposure to MIH will promote restoration of homeostatic BP control, which would be beneficial to participation in daily activities and independence in those with SCI.

DETAILED DESCRIPTION:
Individuals with a spinal cord injury (SCI) above the 6th thoracic vertebrae experience severe autonomic dysfunction. These individuals lose the ability to control blood pressure (BP) during a noxious or non-noxious stimulus below the injury (Autonomic Dysreflexia [AD]) and during positional changes (Orthostatic Hypotension [OH]). The loss of descending autonomic control and subsequent loss of BP control are highly prevalent in individuals with SCI. More importantly, many individuals are unaware of the loss of BP control as most individuals remain asymptomatic. These potentially life-threatening oscillations in BP are known to induce further damage; creating a vicious cycle of continued autonomic and cardiovascular dysfunction which explains the increased cardiovascular related mortality. Unfortunately, there is no effect prophylaxis for autonomic dysfunction in these individuals. Furthermore, the prevalence of sleep disordered breathing (SDB) is high in individuals with SCI (tetraplegia can exceed 90%), and there is no current best clinical practice guidelines for treating SDB in individuals with SCI. The primary treatment is with continuous positive airway pressure (CPAP). Unfortunately, treatment adherence remains poor. Moreover, SDB is known to negatively impact autonomic, cardiovascular, and microvascular function in individuals without SCI. In individuals without an SCI, adherence to CPAP has shown to improve microvascular function. Although no direct evidence is available, individuals with SCI have shown to have a reduction in the frequency of AD when adherent to CPAP suggesting the microvasculature may be a pro-active therapeutic target for AD and OH. Both autonomic dysfunction and SDB are negatively impacted by the lack of motor function following SCI resulting in deconditioning, atrophy of the muscles and vessels, insulin resistance, and reduced metabolic rate. It has been suggested higher CPAP pressure during in-home treatment coupled with increased upper airway resistances are primary physiological barriers to CPAP treatment. Therefore, treatment options that directly improve the blood pressure response to sympathetic activation, upper airway function as well as improve microvascular function are imperative for those with a SCI. The overall goal of the present proposal is to investigate if daily exposure to mild intermittent hypoxia (MIH) can ameliorate autonomic dysfunction in persons with SCI as well as improve mitochondrial and microvascular function. The investigators will recruit individuals with SCI, concurrent SDB, and signs of autonomic dysfunction who will be randomly assign to one of two groups. Treatment will be administered for 8 days over a 2-week period. Both groups will be treated with nightly in-home CPAP over the 8 days. Lastly, individuals will be tested before, and after MIH as well as return to the laboratory 4 weeks later to undergo post-MIH autonomic, cardiovascular, and peripheral muscle function tests. Participants will return 4-weeks later to investigate if there is a sustained impact of therapeutic MIH on autonomic function and SDB. The dissemination of these outcomes could transform the approach to treating autonomic dysfunction and SDB in individuals with SCI. Therefore, this project will determine if MIH combined with CPAP can be used as prophylaxis for autonomic dysfunction in participants with SCI and autonomic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60
2. Motor incomplete spinal cord injury at or above the 12th thoracic vertebrae
3. Signs or symptoms of autonomic dysfunction (this will be determined by the ADFSCI and ISAFSCI questions. The ADFSCI requires a score of 1 on questions 16 and 22, and the ISAFSCI requires a score of 1 on any parameter)
4. Chronic injuries (> 1 year post injury)

Exclusion Criteria:

1. Pregnant
2. Smoker
3. Drug addiction
4. <18 or >60 years of age
5. Complete spinal cord injury
6. Spinal cord injury below the 6th thoracic vertebrae
7. Insulin dependent diabetes
8. Shift workers (ie disrupted circadian rhythm)
9. Active skin breakdown or pressure sores

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Autonomic Dysreflexia | 6 minutes, Pre-Intervention, 1 Day after intervention, 2 weeks after intervention
  Change in systolic blood pressure during dual-thigh occlusion test.

SECONDARY OUTCOMES:
Orthostatic Hypotension | 15 minutes, Pre-Intervention, 1 Day after intervention, 2 weeks after intervention
  The change in systolic blood pressure following positional change (supine to seated)

OTHER OUTCOMES:
Mitochondrial Capacity | 6 minutes, Pre-Intervention, 1 Day after intervention, 2 weeks after intervention
  Oxygen consumption during thigh occlusion
Microvascular function | 6 minutes, Pre-Intervention, 1 Day after intervention, 2 weeks after intervention
  Maximum hyperemic response following 6-minute occlusion test

CONTACTS AND LOCATIONS:
Overall Officials: Gino Panza, PhD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI
Locations (1):
- John D. Dingell VA Medical Center, Detroit, MI, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soltesz AE, Zhao F, Wecht JM, Mateika JH, Panza GS. Mild intermittent hypoxia may improve autonomic dysfunction in persons living with spinal cord injury: a preliminary snapshot. Front Neurosci. 2025 Jul 22;19:1600772. doi: 10.3389/fnins.2025.1600772. eCollection 2025. PMID 40766908